CLINICAL TRIAL: NCT01067794
Title: First-line Treatment of Non-Small Cell Lung Cancer Under Routine Conditions: Observational Study on Overall Survival
Brief Title: Chemotherapy in Treating Patients With Lung Cancer
Acronym: FRAME
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 13095; H3E-EW-B012 (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-02-01; First posted 2010-02-12 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Metastatic; Advanced; Stage IIIB-IV; daily; hospital; practice; setting
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- pemetrexed + platinum: Patients with pemetrexed + platinum doublet, with or without additional targeted agents
  Interventions: Drug: Any platinum-based doublet chemotherapy
- gemcitabine + platinum: Patients with gemcitabine + platinum doublet, with or without additional targeted agents
  Interventions: Drug: Any platinum-based doublet chemotherapy
- taxanes + platinum: Patients with taxanes + platinum doublet, with or without additional targeted agents
  Interventions: Drug: Any platinum-based doublet chemotherapy
- vinorelbine + platinum: Patients with vinorelbine + platinum doublet, with or without additional targeted agents
  Interventions: Drug: Any platinum-based doublet chemotherapy
- others + platinum: Patients with other platinum-based doublet, with or without additional targeted agents
  Interventions: Drug: Any platinum-based doublet chemotherapy

INTERVENTIONS:
Drug: Any platinum-based doublet chemotherapy — Dosage, dosage form, frequency and duration according to daily hospital practice

SUMMARY:
This observational study was planned, with the primary objective to observe patient survival following first-line treatment of patients of Stage IIIB/IV Non-small Cell Lung Cancer (NSCLC) with different platinum-based doublets under routine disease management conditions. Further secondary objectives of this study are to provide insights to what extent histologic subtyping and the use of additional prognostic or predictive biomarkers are currently considered for differential therapeutic decisions under routine conditions. All of these data are critical to evaluate the factors for differential therapeutic decisions and their effect on patient outcomes in a real life setting, and they can only be obtained through observational research.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of non-small cell lung cancer (NSCLC) stage IIIB-IV
* Initiation of first-line treatment for advanced NSCLC with any platinum-based doublet chemotherapy, with or without additional targeted agents
* 18 years of age or older

Exclusion Criteria:

* Participating simultaneously in a study including administration of any investigational drug or procedure at entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (> 18 yrs.) initiating first-line treatment for advanced or metastatic (stage IIIB-IV) NSCLC with any platinum-based doublet chemotherapy, with or without additional targeted agents treated in public hospitals, private hospitals or by office based physicians
Sampling Method: Non-Probability Sample
Enrollment: 1610 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | Treatment start to death from any cause (follow-up assessments until death or until end of study, up to 18 months from Last Patient Entered Treatment)

SECONDARY OUTCOMES:
One-year survival rate | 12 months
Progression-free survival | Treatment start to progression or death (follow-up assessments until death or until end of study, up to 18 months from Last Patient Entered Treatment)
Best tumor response | Treatment start to progression or treatment end

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company

REFERENCES:
- [Derived] Schnabel PA, Smit E, Carpeno Jde C, Lesniewski-Kmak K, Aerts J, Kraaij K, Visseren-Grul C, Dyachkova Y, Taipale K, Girvan A, Moro-Sibilot D. Influence of histology and biomarkers on first-line treatment of advanced non-small cell lung cancer in routine care setting: baseline results of an observational study (FRAME). Lung Cancer. 2012 Dec;78(3):263-9. doi: 10.1016/j.lungcan.2012.09.001. Epub 2012 Oct 4. PMID 23040326